CLINICAL TRIAL: NCT04202185
Title: Evaluation of a Cohort of Congenital Deep Deafness Patients And/or with Auditory Neuropathy, Looking for DFNB9
Acronym: AUDIOFERLINE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190940; 2019-A02968-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Congenital Profound Hearing Loss
Keywords: Auditory neuropathy; DFNB9; Children; Hearing loss; Deafness
MeSH Terms: conditions — Auditory neuropathy; Hearing Loss; Deafness | interventions — Data Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- G1a: infants under 3 years deaf severe to deep
  Interventions: Other: Data collection; Genetic: Genetic analysis
- G1b: children under 16 years of age with audiologically proven auditory neuropathy
  Interventions: Other: Data collection; Genetic: Genetic analysis
- G2: patients <25 years old with one or two Otoferlin mutations
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Retrospective collection data from diagnostic Data collected following to medical exam as part of care
Genetic: Genetic analysis — Research of mutation and identification of genetic panel as part of care
  Groups: G1a; G1b

SUMMARY:
Evaluation of a cohort of deaf children looking for autosomal recessive deafness-9 (DFNB9).

Clinical and audiologic evaluation of patients with known auditive neuropathy / auditory dys-synchrony (ANAD) or recently diagnosed congenital severe to profound hearing loss (HL), and assessing genetic analysis looking for DFNB9. The investigators expect to compile genotypic and phenotypic characterization of 25 children with DFNB9 within 4 years.

DETAILED DESCRIPTION:
ANAD is not a rare type of hearing loss. Nevertheless, its profile is heterogeneous and the pathology remain underdiagnosed. The investigators will screen all new patients with bilateral severe to profound HL, looking for DFNB9. They will analyse their electrophysiology (auditory potential, and otoacoustic emission), and their audio-vestibular profile, at an early stage and one year after inclusion. All patients will be seen in the genetic clinic. Also, the investigators will analyse all patients with ANAD profile and patients known with ANAD.

All informations will provide precise data base to allow a better understanding of the pathology. It might also lead to select the best candidates for future gene therapy

ELIGIBILITY:
G1a / Inclusion Criteria:

* Child from 0 to 3 years old
* Child with severe to profound bilateral deafness newly diagnosed with:
* Average hearing threshold> 70 decibel on each ear
* and / or no response to 70 decibel PEA on each ear
* and / or no response to ASSR

G1b / Inclusion Criteria:

* Child under 16
* Child with newly diagnosed hearing neuropathy : tonal/vocal dissociation (when this is possible), and/or modified PEA, and/or discordant ASSR, and/or OEA present.

G2 / Inclusion Criteria:

* Adult patient under 25 or child
* Patient with deafness with auditory neuropathy
* Patient known to have 1 or 2 mutations of the otoferlin protein

Exclusion Criteria:

* Other type of deafness such as : unilateral deafness, deafness of transmission, malformation syndrome, known genetic familial deafness not DFNB9
* Patient without medical insurance
* Lack of consent to DNA sampling, of one or both biological parents (consent of the care)

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient coming to the Necker Hospital for a deafness visit or for a check-up prior to a cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of deafness caused by DFNB9 | 3 months
  Prevalence and type of bi-allelic pathogenic changes Otoferlin Molecular analysis will be done by Next Generation Sequencing Capture method

SECONDARY OUTCOMES:
Audiological characteristics in free fields at diagnosis | 1 day
  audiometric thresholds on 500, 1000, 2000, 4000 Hz in free fields
Audiological characteristics in separate ears at diagnosis | 1 day
  audiometric thresholds on 500, 1000, 2000, 4000 Hz in separate ears
Audiological characteristics in free fields at 12 months or last record | 12 months
  audiometric thresholds on 500, 1000, 2000, 4000 Hz in free fields
Audiological characteristics in separate ears at 12 months or last record | 12 months
  audiometric thresholds on 500, 1000, 2000, 4000 Hz in separate ears
Electrophysiological characteristics : auditory evoked potentials (PEA) at diagnosis | 1 day
  PEA thresholds per ear
Electrophysiological characteristics : auditory evoked potentials (PEA) at 12 months or last record | 12 months
  PEA thresholds per ear
Electrophysiological characteristics : auditory Steady State Response (ASSR) at diagnosis | 1 day
  ASSR thresholds per ear at 500, 1000, 2000, 4000 Hz
Electrophysiological characteristics : auditory Steady State Response (ASSR) at 12 months or last record | 12 months
  ASSR thresholds per ear at 500, 1000, 2000, 4000 Hz
Electrophysiological characteristics : otoacoustic emissions (OEAs) at diagnosis | 1 day
  OEAs status
Electrophysiological characteristics : otoacoustic emissions (OEAs) at 12 months or last record | 12 months
  OEAs status
Vestibular characteristics : per-oral endoscopic myotomy (PEOM) at diagnosis | 1 day
  PEOM
Vestibular characteristics : per-oral endoscopic myotomy (PEOM) at 12 months or last record | 12 months
  PEOM
Vestibular characteristics : video Head Impulse Test (VHIT) at diagnosis | 1 day
  VHIT
Vestibular characteristics : video Head Impulse Test (VHIT) at 12 months or last record | 12 months
  VHIT
Caloric Tests at diagnosis | 1 day
  Caloric Tests
Caloric Tests at 12 months or last record | 12 months
  Caloric Tests
Clinical development scale at diagnosis | 1 day
  For child under 3 years with : walk age, sitting age and head held age
Clinical development scale at 12 months or last record | 12 months
  For child under 3 years with : walk age, sitting age and head held age

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LOUNDON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Unité d'Audiophonologie et d'Implantation cochléaire - Necker hospital, Paris, France

REFERENCES:
- [Background] Denoyelle F, Petit C. DFNB9. Adv Otorhinolaryngol. 2002;61:142-4. doi: 10.1159/000066822. No abstract available. PMID 12408076
- [Background] Loundon N, Marcolla A, Roux I, Rouillon I, Denoyelle F, Feldmann D, Marlin S, Garabedian EN. Auditory neuropathy or endocochlear hearing loss? Otol Neurotol. 2005 Jul;26(4):748-54. doi: 10.1097/01.mao.0000169044.63970.4a. PMID 16015179
- [Background] Marlin S, Feldmann D, Nguyen Y, Rouillon I, Loundon N, Jonard L, Bonnet C, Couderc R, Garabedian EN, Petit C, Denoyelle F. Temperature-sensitive auditory neuropathy associated with an otoferlin mutation: Deafening fever! Biochem Biophys Res Commun. 2010 Apr 9;394(3):737-42. doi: 10.1016/j.bbrc.2010.03.062. Epub 2010 Mar 16. PMID 20230791
- [Background] Mehl AL, Thomson V. The Colorado newborn hearing screening project, 1992-1999: on the threshold of effective population-based universal newborn hearing screening. Pediatrics. 2002 Jan;109(1):E7. doi: 10.1542/peds.109.1.e7. PMID 11773575
- [Background] Migliosi V, Modamio-Hoybjor S, Moreno-Pelayo MA, Rodriguez-Ballesteros M, Villamar M, Telleria D, Menendez I, Moreno F, Del Castillo I. Q829X, a novel mutation in the gene encoding otoferlin (OTOF), is frequently found in Spanish patients with prelingual non-syndromic hearing loss. J Med Genet. 2002 Jul;39(7):502-6. doi: 10.1136/jmg.39.7.502. No abstract available. PMID 12114484
- [Background] Rouillon I, Marcolla A, Roux I, Marlin S, Feldmann D, Couderc R, Jonard L, Petit C, Denoyelle F, Garabedian EN, Loundon N. Results of cochlear implantation in two children with mutations in the OTOF gene. Int J Pediatr Otorhinolaryngol. 2006 Apr;70(4):689-96. doi: 10.1016/j.ijporl.2005.09.006. Epub 2005 Oct 13. PMID 16226319
- [Background] Roux I, Safieddine S, Nouvian R, Grati M, Simmler MC, Bahloul A, Perfettini I, Le Gall M, Rostaing P, Hamard G, Triller A, Avan P, Moser T, Petit C. Otoferlin, defective in a human deafness form, is essential for exocytosis at the auditory ribbon synapse. Cell. 2006 Oct 20;127(2):277-89. doi: 10.1016/j.cell.2006.08.040. PMID 17055430
- [Background] Varga R, Avenarius MR, Kelley PM, Keats BJ, Berlin CI, Hood LJ, Morlet TG, Brashears SM, Starr A, Cohn ES, Smith RJ, Kimberling WJ. OTOF mutations revealed by genetic analysis of hearing loss families including a potential temperature sensitive auditory neuropathy allele. J Med Genet. 2006 Jul;43(7):576-81. doi: 10.1136/jmg.2005.038612. Epub 2005 Dec 21. PMID 16371502
- [Background] Yasunaga S, Grati M, Cohen-Salmon M, El-Amraoui A, Mustapha M, Salem N, El-Zir E, Loiselet J, Petit C. A mutation in OTOF, encoding otoferlin, a FER-1-like protein, causes DFNB9, a nonsyndromic form of deafness. Nat Genet. 1999 Apr;21(4):363-9. doi: 10.1038/7693. PMID 10192385